CLINICAL TRIAL: NCT00171483
Title: Assessment of the Role of Tegaserod Therapy in the Management of Gastroesophageal Reflux Disease (GERD) Symptoms in Patients With Incomplete Response to Proton Pump Inhibitors (PPIs).
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHTF919BUS30
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2008-01-28 (Estimated); Status verified 2008-01

CONDITIONS: Gastroesophageal Reflux Disease (GERD)
Keywords: GERD; PPI; heartburn; regurgitation
MeSH Terms: conditions — Gastroesophageal Reflux; Heartburn | interventions — tegaserod

INTERVENTIONS:
Drug: Tegaserod

SUMMARY:
Study to assess the effects of tegaserod added to PPI therapy in the resolution of heartburn and regurgitation in patients with incomplete relief from PPIs .

ELIGIBILITY:
Inclusion Criteria:

* Heartburn for at least 3 days in the week prior to screening
* Regurgitation for at least 3 days in the week prior to screening
* Stable dose PPI therapy > 4 weeks
* Incomplete relief on daily PPI therapy > 4 weeks

Exclusion Criteria:

* Evidence of structural abnormality of the gastrointestinal tract or disease/conditions
* Previous gastrointestinal surgery that may influence esophageal motor function
* Evidence of cathartic colon or a history of laxative use

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2004-01; Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
To determine the effect of 6 weeks of tegaserod in addition to proton pump inhibitors on heartburn and regurgitation (weekly assessment)

SECONDARY OUTCOMES:
To evaluate the sensitivity of three global symptom assessments of GERD related to complaints (end of treatment compared to baseline)
To evaluate frequency, severity and bothersomeness of individual GERD symptoms (daily assessments)
To assess baseline characteristics that may predict a positive response to tegaserod add-on therapy in GERD patients
To assess patient satisfaction with treatment (end of treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis
Locations (7):
- United States (7):
  - Consultants for Clinical Research of South Florida, Boynton Beach, Florida
  - Miami Research Associates, Miami, Florida
  - University Clinical Research, Pembroke Pines, Florida
  - Department of Internal Medicine - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - Consultants for Clinical Research, Cincinnati, Ohio
  - Metropolitan Research, Fairfax, Virginia
  - The Wisconsin Center for Advanced Research, Milwaukee, Wisconsin